CLINICAL TRIAL: NCT06011577
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of REL-1017 as an Adjunctive Treatment for Major Depressive Disorder (RELIGHT)
Brief Title: Randomized, Double-Blind, Placebo-Controlled Trial of REL-1017 as Adjunctive Treatment for MDD
Acronym: RELIGHT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Program Discontinued
Sponsor: Levomecor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REL-1017-304
Expanded Access: NCT06009003 (Temporarily not available)
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Depression
Keywords: REL-1017; esmethadone; Relmada; antidepressant; adjunctive; NMDA receptor antagonist; Relight; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REL-1017 25 mg (Experimental): During the double blind treatment period (28 days), participants will take 1 tablet of REL-1017 25 mg, orally, per day in addition to their ongoing antidepressant (ADT)
  Interventions: Drug: REL-1017
- Placebo (Placebo Comparator): During the double blind treatment period (28 days), participants will take 1 tablet of placebo, orally, per day in addition to their ongoing antidepressant (ADT)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REL-1017 — REL-1017 tablet
  Other Names: esmethadone
  Arms: REL-1017 25 mg
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
A Phase 3, randomized, double-blind, placebo-controlled, multicenter trial of REL-1017 in patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
This is an outpatient, 2-arm, Phase 3, multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of REL-1017 once daily (QD) as an adjunctive treatment of Major Depressive Disorder in patients with inadequate response to ongoing background antidepressant treatment. Eligible patients will continue to take their background antidepressant therapy and be randomized in a 1:1 ratio to treatment with REL-1017 or placebo for a 4 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 35.0 kg/m2.
* Diagnosed with Major Depressive Disorder (MDD) based on Structured Clinical Interview for DSM-5 (SCID-5) for MDD.
* Inadequate response to 1 to 3 adequate antidepressant treatments in the current MDE.

Exclusion Criteria:

* Psychiatric hospitalization during the current major depressive episode.
* History or presence of clinically significant health conditions which in the opinion of the Investigator would negatively impact the safety of the participant.
* Participants who, in the Investigator's judgment, are at significant risk for suicide.
* Pregnant or planning to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in MADRS Total Score From Baseline to Day 28 | Day 28
  The MADRS is a 10-item scale and items are scored between 0-6 points. For each item, a score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity. A maximum total score is 60 points.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Greene, PhD, Study Director — Relmada Therapeutics
Locations (35):
- United States (35):
  - Relmada Site, Dothan, Alabama
  - Relmada Site, Homewood, Alabama
  - Relmada Site, Anaheim, California
  - Relmada Site, Lafayette, California
  - Relmada Site, Newport Beach, California
  - Relmada Site, Orange, California
  - Relmada Site, Redlands, California
  - Relmada Site, Sherman Oaks, California
  - Relmada Site, Farmington, Connecticut
  - Relmada Site, Brandon, Florida
  - Relmada Site, Hialeah, Florida
  - Relmada Site, Jacksonville, Florida
  - Relmada Site, Miami, Florida
  - Relmada Site, Okeechobee, Florida
  - Relmada Site, Tampa, Florida
  - Relmada Site, Springfield, Illinois
  - Relmada Site, Baltimore, Maryland
  - Relmada Site, Mankato, Minnesota
  - Relmada Site, Toms River, New Jersey
  - Relmada Site, Brooklyn, New York
  - Relmada Site, Cedarhurst, New York
  - Relmada Site, New York, New York
  - Relmada Site, Philadelphia, Pennsylvania
  - Relmada Site, Franklin, Tennessee
  - Relmada Site, Memphis, Tennessee
  - Relmada Site, Austin, Texas
  - Relmada Site, Bellaire, Texas
  - Relmada Site, Friendswood, Texas
  - Relmada Site, Houston, Texas
  - Relmada Site, Wichita Falls, Texas
  - Relmada Site, Clinton, Utah
  - Relmada Site, Draper, Utah
  - Relmada Site, Rutland, Vermont
  - Relmada Site, Charlottesville, Virginia
  - Relmada Site, Seattle, Washington

REFERENCES:
- See also: Study Homepage — http://www.relightstudies.com